CLINICAL TRIAL: NCT00772044
Title: Randomized, Double-blind Study to Compare Safety and Effectiveness of the ProventTM Professional Sleep Apnea Therapy Device to Sham for the Non-invasive Treatment of OSAH
Brief Title: Randomized Study of Provent Versus Sham Device to Treat Obstructive Sleep Apnea
Acronym: AERO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ventus Medical, Inc. (Industry)
Responsible Party: Connie Rey, Director, Clinical Affairs, Ventus Medical, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C009
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Obstructive Sleep Apnea Hypopnea; OSA; OSAH
Keywords: OSA; sleep apnea; apnea; AHI
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provent (Active Comparator): Those receiving the active device
  Interventions: Device: Provent Professional Sleep Apnea Therapy Device
- Sham (Sham Comparator): Those receiving sham device
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Provent Professional Sleep Apnea Therapy Device — Application of active device (Provent)
  Other Names: Provent
  Arms: Provent
Device: Sham Device — Sham device will be applied
  Arms: Sham

SUMMARY:
Primary Endpoints:

•Comparison of difference in AHI at one-week in-lab polysomnography between "device on" and "device off" nights, controlling for sleep position (supine vs. non-supine)

Secondary Endpoints: By polysomnography, reduction in:

* AHI with device on vs. off at 3 months, controlling for sleep position
* Oxygen desaturation index with device on vs. off
* Arousal index with device on vs. off
* Duration of snoring with device on vs. off
* Epworth Sleepiness Scale

Patient acceptance, in terms of:

* Refusal rate at screening
* Discontinuation rate during follow-up
* Daily compliance rate
* Device-related adverse events
* Serious adverse events

DETAILED DESCRIPTION:
Please see summary above

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis of OSA
3. AHI > 10 on diagnostic PSG performed within last 3 months
4. Investigator believes that subject can benefit from OSA tx
5. Subject understands and is willing and able to comply with study requirements

Exclusion Criteria:

1. Use of any device that interferes with nasal/oral breathing
2. Persistent blockage of one or both nostrils
3. Any chronic sores or lesions on the inside/outside of the nose
4. Chronic use of nasal decongestants other than nasal steroids
5. Oxygen saturation < 75% for > 10% of the diag. PSG
6. Oxygen saturation < 75% for > 25% of the first 4 hours of the diag. PSG
7. Prior or near-miss motor vehicle accident due to sleepiness (last 12 mo.)
8. Current use of hypnotics, anxiolytics, sedating antidepressants, anticonvulsants, sedating antihistamines, stimulants, or other medications likely to affect neurocognitive function and/or alertness
9. History of allergic reaction to acrylic-based adhesives
10. Current acute upper respiratory inflammation/infection or perforation of the tympanic membrane
11. History of frequent and/or poorly treated severe nasal allergies or sinusitis
12. Narcolepsy, idiopathic hypersomnolence, chronic insomnia, RLS, REM sleep behavior disorder or any other diagnosed or suspected sleep disorder
13. Current use of diurnal or nocturnal supplemental oxygen
14. History of CPAP use in the home for OSA tx
15. History of use of oral appliances for OSA tx
16. History of prior surgery for OSA
17. Currently working night or rotating shifts
18. Consumption of > 10 caffeinated beverages per day
19. History of severe cardiovasc. disease, including NYHA Class III or IV heart failure, CAD with angina or MI/stroke in past 6 months
20. History of cardiac rhythm disturbance
21. Uncontrolled hypertension (SBP > 180 or DBP > 105 mm Hg)
22. Uncontrolled hypotension(SBP < 80 or DBP < 55 mm Hg
23. History of severe respiratory disorders or unstable respiratory disease
24. Any other serious, uncontrolled medical condition
25. Females of child bearing age who are pregnant or intending to become pregnant
26. Consumes more than 3 drinks of alcohol/day
27. Chronic neurologic disorders
28. Cancer, unless in remission for more than 1 year
29. Current psychiatric illness
30. Smokers whose habit interferes with the overnight PSG
31. Any known illicit drug usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of difference in AHI at one-week in-lab polysomnography between "device on" and "device off" nights, controlling for sleep position (supine vs. non-supine) | 3 months

SECONDARY OUTCOMES:
Reduction in AHI, Oxygen desat index, Arousal index & Duration of snoring w/ device on/off;ESS,Patient acceptance,Device-related AEs & SAEs | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Berry, M.D., Principal Investigator — University of Florida; Connie A Rey, Study Director — Ventus Medical
Locations (17):
- United States (17):
  - Pulmonary Associates, Glendale, Arizona
  - Pulmonary Associates, Phoenix, Arizona
  - Stanford Center for Human Sleep Research, Redwood City, California
  - Gaylord Sleep Medicine, Wallingford, Connecticut
  - University Of Florida College of Medicine, Gainesville, Florida
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Chicago Sleep Group of Suburban Lung Associates, Elk Grove Village, Illinois
  - Kentucky Research Group, Louisville, Kentucky
  - Sleep Health Center, Brighton, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Sleep Medicine and Research Center, Chesterfield, Missouri
  - The Corvallis Clinic, Corvallis, Oregon
  - SleepMed of South Carolina, Columbia, South Carolina
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Berry RB, Kryger MH, Massie CA. A novel nasal expiratory positive airway pressure (EPAP) device for the treatment of obstructive sleep apnea: a randomized controlled trial. Sleep. 2011 Apr 1;34(4):479-85. doi: 10.1093/sleep/34.4.479. PMID 21461326